CLINICAL TRIAL: NCT02923011
Title: Phase III Study to Compare the Effectiveness of Magnetic Resonance Guided Focused Ultrasound With Computed Tomography Guided Radiofrequency Ablation for Treatment of Osteoid Osteomas
Brief Title: Comparative Effectiveness of MRgFUS Versus CTgRFA for Osteoid Osteomas
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Matthew Bucknor (Other)
Collaborators: Focused Ultrasound Foundation (Other)
Responsible Party: Sponsor-Investigator, Matthew Bucknor, Assistant Professor in Residence, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUS513
Record Dates: First submitted 2016-09-30; First posted 2016-10-04 (Estimated); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Osteoid Osteoma
MeSH Terms: conditions — Osteoma, Osteoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- MRgFUS (Active Comparator): Magnetic resonance-guided focused ultrasound ablation
  Interventions: Device: MRgFUS
- CTgRFA (Active Comparator): Computed tomography-guided radiofrequency ablation
  Interventions: Device: CTgRFA

INTERVENTIONS:
Device: MRgFUS — Magnetic resonance-guided focused ultrasound ablation of osteoid osteoma
  Arms: MRgFUS
Device: CTgRFA — Computed tomography-guided radiofrequency ablation of osteoid osteoma
  Arms: CTgRFA

SUMMARY:
Osteoid osteomas are painful, benign bone tumors that occur most frequently in young males between ages 10 and 20 years. The goal of the proposed study is based on the premise that MRgFUS is noninferior to CT-guided radiofrequency ablation (CTgRFA), in terms of pain reduction following treatment of osteoid osteomas, and offers possible improvements with regards to 1) post-procedural pain, 2) clinical resource utilization, 3) patient experience, and/or 4) adverse events. The data from the current study would provide clinicians important information in deciding between treatment options for ablation of osteoid osteomas.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ages ≥ 8 years old.
2. Diagnosis of osteoid osteoma as confirmed when a musculoskeletal radiologist and orthopedic oncologist agree that a patient's imaging and clinical history are most compatible with the diagnosis of osteoid osteoma. A patient referred by a clinician other than orthopedic oncologist will require a clinic visit with an orthopedic oncologist for study inclusion.
3. Patients must have medically uncontrolled pain from an osteoid osteoma, as defined by pain, which, in the view of the referring orthopedic oncologist significantly interferes with that patient's activities of daily living. Pain may be refractory to management with medications because of inadequate pain control, or because of side effects of the pain medication.
4. If patients have an additional site of pain, it must be 2 points less severe and distinguishable from the pain at the osteoid osteoma site.
5. Patients (or guardians/parents) who are able and willing to give consent (or assent where applicable) and able to attend all study visits.
6. No prior interventional therapy for the osteoid osteoma.
7. Able to safely undergo MRI exam, tolerate being in an MRI scanner, and receive anesthesia/sedation for the treatment.
8. Targeted bone/tumor interface is accessible to the ExAblate device and located in a rib, extremity (excluding intra-articular location), pelvis, shoulders (including clavicles), or the sternum.
9. Targeted lesion must be deeper than 1 cm from the skin.
10. Targeted lesion must be clearly visible by non-contrast MRI.
11. Karnofsky Performance Status > 60.

Exclusion Criteria:

1. Patients a) who need surgical stabilization of the affected bone (elevated fracture risk) or b) whose targeted tumor is at an impending fracture site, as determined by the referring orthopedic oncologist.
2. Targeted tumor in the skull/spine.
3. Targeted tumor is < 1 cm from a major nerve.
4. Pregnancy.
5. Patients with an acute medical condition (e.g. pneumonia, sepsis) that is expected to hinder them from completing this study.
6. Patients with unstable cardiac status including: patients on anti-arrhythmic drugs, unstable angina pectoris, documented myocardial infarction within six months of protocol entry, congestive heart failure requiring medication (other than diuretic).
7. Severe hypertension (diastolic BP > 100 on medication)
8. Patients with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices.
9. Patients with an active infection or severe hematological, neurological, or other uncontrolled disease.
10. Severe cerebrovascular disease.
11. Known intolerance or allergy to medications used for sedation/anesthesia.
12. Known intolerance or allergy to MR contrast agent (gadolinium chelates).
13. Patients unable to communicate with the investigator and staff.
14. Patients with persistent pain undistinguishable from the target lesion.

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2017-03-28 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of resolution of pain (worst visual analog scale score over last 24 hours < 2.0) | 1 month
  1 month after treatment, worst VAS score over the last 24 hours will be assessed

SECONDARY OUTCOMES:
Procedure time | Treatment day
  On the day of the treatment, the procedure time will be recorded
Patient preference | 2 weeks
  2 weeks after treatment, patient preference surveys will be assessed
Patient quality of life | 1 month
  1 month after treatment, patient quality of life surveys will be assessed
Medication use | 5 days before, five days after, 1 month after
  Self reported medication use for 5 days before, five days after, and 1 month after the treatment
Adverse events | 1 month
  All adverse events occurring within the first month will be recorded at 1 month following the procedure
Worst VAS | First 5 days, 1 week, 2 weeks, 3 weeks, 1 month, 6 months, 12 months
  Worst VAS over the last 24 hours will be assessed for each of the first 5 days following the treatment and then at 1 week, 2 weeks, 3 weeks, 1 month, 6 months, and 12 months following the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Bucknor, MD, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - Stanford Medical Center, Palo Alto, California
  - UCSF Imaging Center, San Francisco, California
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No